CLINICAL TRIAL: NCT04338334
Title: Effectiveness of Cohesive Bandage on Axillary Web Syndrome After Breast Cancer Surgery: a Randomized Controlled Trial
Brief Title: Effectiveness of Cohesive Bandage on Axillary Web Syndrome After
Acronym: CBaws
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Principal investigator & Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OE20/2020
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Axillary Web Syndrome
Keywords: Cohesive bandage; Physical Therapy; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (Active Comparator): Control group includes physical therapy protocol composed of manual lymph-drainage technique in axilla, and proximal ipsilateral arm, specific thumb manual lymph-drainage on the taut cords to make them gradually more flexible, in conjunction with progressive active arm therapeutic exercises.
  Interventions: Other: Manual drainage & arm therapeutic exercise
- COHESIVE BANDAGE GROUP (Experimental): Cohesive bandage is a self-adherent lightweight bandage, made of a porous nonwoven polyester material. A single self-adherent inelastic bandage will be directly applied at full stretch on cleaned and dried skin (10cm 3M CobanTM Minnesota Mining and Manufacturing Co, United States) in a spiral method around the limb, starting at the hand and a layer overlap of 50%, so that the greatest compression was located at the distal points, gradually decreasing toward the proximal shoulder part. Cohesive latex-free bandages will be available for those allergic women. Women will do progressive active arm therapeutic exercises with bandaging.
  Interventions: Other: Cohesive bandaging & arm therapeutic exercise

INTERVENTIONS:
Other: Manual drainage & arm therapeutic exercise — See arm/group descriptions.
  Arms: CONTROL GROUP
Other: Cohesive bandaging & arm therapeutic exercise — See arm/group descriptions.
  Arms: COHESIVE BANDAGE GROUP

SUMMARY:
Objective: To determine the effectiveness of cohesive bandage on the axillary web syndrome in improving pain, reducing swelling and increasing mobility and functionality of the shoulder. Design: randomized single-blinded controlled trial. Follow-up: five physical therapy assessments: pre-intervention; post-intervention, 3 and 6 months post-intervention post-intervention. Participants: 90 consecutive women diagnosed with axillary web syndrome after undergoing unilateral breast cancer surgery with ALND or SLND at the Prıíncipe de Asturias Hospital in Alcalà de Henares, Madrid (Spain). Randomization: women will be randomly assigned to two groups by EpiData 3.1 software. Interventions: Control group: Physical Therapy composed of manual lymph-drainage technique in axilla, and proximal ipsilateral arm, specific thumb manual lymph-drainage on the taut cords to make them gradually more flexible, in conjunction with progressive active arm therapeutic exercises; Intervention group: progressive active arm therapeutic exercises with cohesive bandage.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral breast cancer;
* Breast surgery with lymphadenectomy and / or sentinel lymph node biopsy;
* Axillary web syndrome in upper limb of the operated side;
* Consent to participate in the study;
* No contraindications.

Exclusion Criteria:

* Cognitive impairment;
* Visual impairment for reading;
* Lymphedema;
* Bilateral breast cancer;
* Systemic disease (metastases),
* Infection;
* Locoregional recurrence.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Subjective pain | 4 assessments to evaluate change from baseline: at baseline, after the intervention period (6 weeks from baseline), 3 and 6 months after the intervention.
  Visual Analogue Scale (0-10 cm)

SECONDARY OUTCOMES:
Change from baseline in Range of shoulder motion | 4 assessments to evaluate change from baseline: at baseline, and after the intervention period (6 weeks from baseline), 3 months and 6 months after the intervention.
  Inclinometer (measured in grades)
Change from baseline in perceived shoulder disability | 4 assessments to evaluate change from baseline: at baseline, and after the intervention period (6 weeks from baseline), 3 months and 6 months after the intervention.
  Oxford Shoulder Score. The OSS is a unidimensional score comprising 12 questions about pain and disability involving activities of daily routine. Thus, each of the 12 questions is scored from 0 to 4, with 4 representing best outcome/least symptoms. Scores from each question are summed so the overall score run from 0 to 48 with 48 being the best outcome; so that the lower scores indicate more pain and disability. The OSS Spanish version is applicable, reliable, valid, and responsive to assess shoulder disability in Spanish women after breast cancer treatment
Change from baseline in QoL | 4 assessments to evaluate change from baseline: at baseline, and after the intervention period (6 weeks from baseline), 3 months and 6 months after the intervention.
  FACTB+4. Health-related quality of life (HRQoL): HRQoL was measured with the Functional Assessment of Cancer Therapy-Breast (FACT-B) Spanish version 4. FACT-Bv4 is a 40-item questionnaire designed to measure multidimensional HRQoL in women with breast cancer. The 40 items cover four generic scales of well-being (Physical, Emotional, Social, and Functional) and two side-specific subscales: Breast Cancer (9 items) and Arm (4 items). The Arm-specific subscale assesses arm morbidity: 1) pain, 2) poor range of arm movements, 3) numbness, and 4) stiffness. The Breast Cancer subscale plus the arm subscale range from 0 to 56 points. The Trial Outcome Index (TOI) is the sum of Physical and Functional wellbeing plus Breast Cancer Subscale (range 0-92 points). The FACT-B total score can range from 0 to 144, with a higher score indicating better HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: María Torres-Lacomba, PhD, Principal Investigator — University of Alcalá
Locations (1):
- María Torres-Lacomba, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No